CLINICAL TRIAL: NCT02567773
Title: A Randomized Double-blind (Sponsor Unblind) Placebo Controlled Study in Healthy Subjects to Evaluate: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Repeat Doses of GSK2881078, the Selective Androgen Receptor Modulator With an Open Label Dosing Arm to Evaluate the Effect of CYP3A4 Inhibition on Pharmacokinetics of GSK2881078
Brief Title: Safety, Tolerability, Pharmacokinetic (PK), and Pharmacodynamic Study of GSK2881078 and Study to Evaluate the Effect of CYP3A4 Inhibition on PK of GSK2881078
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 204699
Record Dates: First submitted 2015-09-03; First posted 2015-10-05 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Cachexia
Keywords: Itraconazole; GSK2881078; CYP3A4; Selective Androgen Receptor Modulator; Safety; Pharmacokinetics; Tolerability
MeSH Terms: conditions — Cachexia | interventions — GSK2881078; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: GSK2881078 (Experimental): The first cohort subjects will receive GSK2881078 1.5 mg (for males) or 0.75 mg (for females) twice daily for 3 days followed by once daily for 25 days. The subsequent cohort subjects will receive GSK2881078 doses selected after reviewing the unblinded data from at least 2 weeks of dosing of at least 6 subjects in the first cohort. Each cohort subjects will receive GSK2881078 dose twice daily for the first 3 days followed by 25 days of once daily.
  Interventions: Drug: GSK2881078
- Part A: Placebo (Placebo Comparator): Subjects will receive placebo twice daily for 3 days followed by once daily for 25 days.
  Interventions: Drug: Placebo
- Part B: GSK2881078-Itraconazole (Experimental): Subjects will receive GSK2881078 (dose level will be determined based on the results from Part A) on Day 1 of Period-1 and Day 6 of Period-2. Subjects will also receive itraconazole 200 mg twice daily on Day1 of Period-2 and 200 mg once daily on Days 2-34 of Period-2.
  Interventions: Drug: GSK2881078; Drug: Itraconazole

INTERVENTIONS:
Drug: GSK2881078 — GSK2881078 hot melt solutions, ranging in concentration from 0.05 mg/g to 50 mg/g, will be prepared by weighing drug substance directly into specific quantities of the hot melt vehicle solution. Subjects will be administered GSK2881078 (dose for Cohort 1: 0.75 mg for females and 1.5 mg for males) hot melt solution within capsule orally with water.
  Arms: Part A: GSK2881078; Part B: GSK2881078-Itraconazole
Drug: Placebo — Subjects will be administered as hot melt vehicle placebo within capsule orally with water.
  Arms: Part A: Placebo
Drug: Itraconazole — Subjects will be administered as two capsules of itraconazole 100 mg (200 mg) orally with water.
  Arms: Part B: GSK2881078-Itraconazole

SUMMARY:
GSK2881078 is a selective androgen receptor modulator (SARM) that is being evaluated for effects on muscle growth and strength in subjects with muscle wasting to improve their physical function. Part A of this study will evaluate the safety, efficacy and pharmacokinetics of GSK2881078 in healthy, older men and post-menopausal women who will take daily dosing for 28 days and be followed for a total of 70 days. Part B of this study will characterize the effect of Cytochrome P450 3A4 (CYP3A4) inhibition on the GSK2881078 pharmacokinetics. Part B will only be conducted if safe and efficacious dose is identified in Part A. Part A will include healthy older males and post-menopausal females; and randomize approximately 60 subjects (about 15 per cohort [4 cohorts]) to complete approximately 48 (about 12 per cohort). Part B will enroll one cohort of approximately 15 healthy male subjects to complete approximately 12. The study duration will be approximately 115 days for Part A and 122 days for Part B.

ELIGIBILITY:
Inclusion Criteria:

* Age: Part A: Between 50 and 75 years of age inclusive, at the time of signing the informed consent form. Part B: Between 18 and 60 years of age inclusive, at the time of signing the informed consent form.
* Healthy as determined by the investigator. Subjects with hypertension, hyperlipidemia or hypothyroidism, well controlled and stable on a single medication, may also be included.
* Subject values for Hemoglobin (Hgb) must be within the normal range (plus or minus 10%).
* Estimated glomerular filtration rate (GFR) >=60 milliliter (mL)/minute (min)/1.73 square meter (m^2).
* Body Mass Index (BMI) within the range 19 - 32 kilogram (kg)/m^2 (inclusive).
* Sex: Part A: Male or Female; Part B: Male Males: Male subjects with female partners of child bearing potential must agree to use a condom from the time of first dose of study medication until the final follow-up visit.

Females: A female subject is eligible to participate if she is post-menopausal.

Exclusion Criteria:

* Alanine transaminase (ALT) and bilirubin >1.1x upper limit of normal (ULN) (isolated bilirubin >1.1xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease including fatty liver, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) > 450 msec. Heart rate: <40 and >100 beats per minute, PR Interval: <120 and >210 millisecond (msec), QRS duration: <70 and >120 msec.
* Subjects with a history at any time in the past of coronary artery disease, congestive heart failure, angina, myocardial infarction, any cardiac surgery, valvular heart disease, clinically significant arrhythmia, dyspnea, pulmonary edema, stroke, or transient ischemic attack.
* Subjects with a history of clinically significant endocrine, gastrointestinal, hepatic, cardiovascular, neurological, haematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
* Subjects with a history of malignancy that is not in complete remission for at least 5 years or 1 year for non-melanoma skin carcinoma.
* Male subjects with a family history of early onset (55 years of age or younger) prostate cancer or 2 or more direct family members with prostate cancer.
* Unable to refrain from prescription or non-prescription drugs as described in protocol.
* History of regular alcohol consumption within 6 months of the study.
* History of drug or alcohol abuse within 5 years prior to the Screening Period.
* Unable to refrain from consumption (whole fruit or juice) of seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, or grapefruit hybrids.
* Regular, strenuous exercise or weightlifting >2 times per week for at least 2 weeks prior to screening visit or intent to start a new exercise routine during the study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof.
* Metal implants (contraindicated for MRI and disrupt DXA imaging). These include intra-orbital metal fragments.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). Subjects who previously received GSK2881078 are allowed to participate in this trial, with the same timeline restrictions.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Prostate Specific Antigen (PSA) >4.0 nanograms (ng)/mL.
* High-density lipoprotein cholesterol (HDL-C) <35 milligram (mg)/deciliter (dL).
* Thyroid stimulating hormone (TSH) >10 mIU/L, test may be repeated or thyroid panel discussed with Medical Monitor.
* Testosterone < 0.9 lower limit of normal range (LLNR) - 10%, test may be repeated, or free testosterone determined also <0.9 LLNR.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Part A: Blood pressure as a measure of safety and tolerability | Up to Day 70
  Blood pressure will be recorded whilst the subject is in a semi -supine position, having rested in this position for at least 10 minutes.
Part A: Heart rate as a measure of safety and tolerability | Up to Day 70
  Heart rate will be recorded whilst the subject is in a semi -supine position, having rested in this position for at least 10 minutes.
Part A: Cardiac telemetry as a measure of safety and tolerability | Up to Day 28
  Continuous cardiac telemetry will be performed for at least 8 hours post-dose.
Part A: Electrocardiogram (ECG) as a measure of safety and tolerability | Up to Day 70
  Triplicate or single 12-lead ECGs will be obtained at each timepoint and will be recorded whilst the subject is in a semi-supine position, having rested in this position for at least 10 minutes.
Part A: Composite of clinical laboratory parameters including hematology, clinical chemistry, and lipid blood panel (fasting) as a measure of safety and tolerability | Up to Day 70
Part A: Number of subjects with adverse events (AEs) | Up to Day 70
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Part A: area under the plasma drug concentration curve from time zero to the time of last quantifiable concentration (AUC0-t) for GSK2881078 after 14 and 28 days of dosing | Day 14-15 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and Day 28-30 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24 36, and 48 hours post-dose)
Part A: area under the plasma drug concentration curve from time zero to end of dosing interval (AUC0-tau) for GSK2881078 after 14 and 28 days of dosing | Day 14-15 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and Day 28-30 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24 36, and 48 hours post-dose)
Part A: maximum observed plasma drug concentration (Cmax) for GSK2881078 after 14 and 28 days of dosing | Day 14-15 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and Day 28-30 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24 36, and 48 hours post-dose)
Part A: time to maximum observed plasma drug concentration (Tmax) for GSK2881078 after 14 and 28 days of dosing | Day 14-15 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and Day 28-30 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24 36, and 48 hours post-dose)
Part A: terminal half-life (t1/2) for GSK2881078 after 14 and 28 days of dosing | Day 14-15 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and Day 28-30 (Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24 36, and 48 hours post-dose)
Part B: area under the plasma drug concentration curve from time zero to infinity (AUC0- infinity) of GSK2881078 in absence and presence of itraconazole | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 336, 504 and 672 hours post dose in both periods
Part B: Cmax of GSK2881078 in absence and presence of itraconazole | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 336, 504 and 672 hours post dose in both periods

SECONDARY OUTCOMES:
Part A: Change from baseline in appendicular mass as assessed by Dual-energy X-ray Absorptiometry (DXA) | Baseline and up to Day 70
  Appendicular lean mass will be calculated from the regional lean mass measurements of the arms and legs.
Part A: Change from baseline in total lean mass as assessed by DXA | Baseline and up to Day 70
  Output from DXA will be used to measure total lean mass.
Part A: Change from baseline in thigh muscle volume as assessed by MRI | Baseline and up to Day 70
  MRI cross-sectional thigh scans will be performed for each cohort in Part A of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States